CLINICAL TRIAL: NCT02382393
Title: Reliability and Validity of Online Cognitive Assessments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumos Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: LL002(p)
Record Dates: First submitted 2015-03-03; First posted 2015-03-06 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Volunteers
Keywords: cognitive assessment; Brain Performance Test; Lumosity; concurrent validity; computerized assessment

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BPT, Computerized Assessment (Experimental): Participants will first take the Brain Performance Test (BPT) and then a third party validated assessment battery.
  Interventions: Other: Brain Performance Test (BPT, Lumos Labs, Inc); Other: Computerized Assessment
- Computerized Assessment, BPT (Experimental): Participants will take a third party validated assessment battery and then the Brain Performance Test (BPT).
  Interventions: Other: Brain Performance Test (BPT, Lumos Labs, Inc); Other: Computerized Assessment

INTERVENTIONS:
Other: Brain Performance Test (BPT, Lumos Labs, Inc) — A brief, repeatable, online battery of cognitive assessments used to measure functioning in five cognitive domains across time.
Other: Computerized Assessment — a validated, computerized cognitive assessment tool

SUMMARY:
The purpose of this study is to evaluate the concurrent validity (correlation coefficient of scores at 1 time point) between the Brain Performance Test (BPT, Lumos Labs, Inc.) and a validated third party computerized assessment.

DETAILED DESCRIPTION:
Each subject will complete two sessions, each approximately 1 hour in total duration, approximately 2 weeks apart for a total duration of participation of 2 hours over 2 weeks

ELIGIBILITY:
Inclusion Criteria:

* Electronically signed informed consent
* 18 years of age or older
* Native English-Speaker
* Consistent access to a computer with stable internet connection

Exclusion Criteria:

* Under 18 years of age
* Native language other than English
* Visual impairment that impedes computer use
* Has taken a cognitive assessment or done cognitive training in the past year

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1152 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
BPT Grand Index Score at Time 1 | Baseline
Computerized Assessment Index at Time 1 | Baseline
Selected raw and scaled BPT and Computerized Assessment matched subtest scores at Time 1 | Baseline

SECONDARY OUTCOMES:
BPT Grand Index at Time 1 and Time 2 | Baseline to 2 weeks
Computerized Assessment Index at Time 1 and Time 2 | Baseline to 2 weeks
Raw and scaled BPT subtest scores at Time 1 and Time 2 | Baseline to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Morrison, PhD, Principal Investigator — Lumos Labs, Inc.
Locations (1):
- Lumos Labs, Inc., San Francisco, California, United States

REFERENCES:
- See also: Click here for more information about joining this study. — https://lumosity.com/landing?refer=8838